CLINICAL TRIAL: NCT05283876
Title: Excimer Light Effect on Neurogenic Inflammation in Developing Versus Stationary Psoriasis Lesions
Brief Title: Excimer Light in Psoriasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa Salah El-Din El-Mesidy, Dr., Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Excimer light in psoriasis
Record Dates: First submitted 2022-02-17; First posted 2022-03-17 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active psoriasis (Active Comparator)
  Interventions: Device: Excimer light
- Stable psoriasis (Active Comparator)
  Interventions: Device: Excimer light

INTERVENTIONS:
Device: Excimer light — Excimer light sessions

SUMMARY:
The aim of this study is to determine the standard tissue levels of SP and its receptor in lesional skin of psoriasis patients in both developing and stationary stages before and after excimer light therapy.

ELIGIBILITY:
Inclusion Criteria:

* Type of Psoriasis: plaque psoriasis.
* Less than 10% surface area.

Exclusion Criteria:

* Erythrodermic psoriasis
* Pustular psoriasis
* Topical treatment for psoriasis for the past 2 weeks.
* Systemic retinoids in the last 2 years.
* Systemic treatments (including any drugs that affect SP level as Aprepitant) in the last 3 months.
* Contraindications to excimer light therapy (history of skin malignancy or precancerous conditions like xeroderma pigmentosum or photosensitivity)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Excimer laser efficiency in active and stable psoriasis | through study completion, an average of 6 months
  Determine the clinical improvement using Local psoriasis severity index
Excimer laser efficiency on neurogenic inflammation | through study completion, an average of 6 months
  level of affection of the neurogenic inflammation in psoriasis lesions after using Excimer light therapy. Determine substance P and its receptor levels before and after therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Al Ainy Faculty of medicine, Cairo, Egypt